CLINICAL TRIAL: NCT01835626
Title: A Phase II Study of Radiation Therapy and Vismodegib, for the Treatment of Locally Advanced Basal Cell Carcinoma of the Head and Neck
Brief Title: Phase II Study of Radiation Therapy and Vismodegib for Advanced Head/Neck Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sue Yom (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sue Yom, Associate Professor, Department of Radiation Oncology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122011; NCI-2013-00871 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-04-10; First posted 2013-04-19 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Locally Advanced Basal Cell Carcinoma; Skin Cancer; Cutaneous Malignancy
Keywords: Locally advanced basal cell carcinoma; Skin cancer; Radiation therapy; Vismodegib; Head and neck cancer; Cutaneous malignancy
MeSH Terms: conditions — Skin Neoplasms; Head and Neck Neoplasms | interventions — HhAntag691; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib and Radiation Therapy (Experimental): 150mg Vismodegib will be taken once a day, daily. Radiation therapy will be started after the patient has completed taking vismodegib for 12 weeks. The patient will take daily vismodegib through the completion of radiation therapy. The patient will receive radiation once a day, Monday through Friday, for 7 weeks. Each radiation treatment may take up to 30 minutes.
  Interventions: Drug: Vismodegib; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Vismodegib — Vismodegib will be taken daily for 12 weeks. It should be taken at approximately the same time each day. Patients will be given a supply of vismodegib on Week 1, Day 1 to last until their next study visit. They will be asked to keep a record of each dose of vismodegib you take. After 12 weeks, they will be evaluated again to make sure they are still eligible to participate in the study. If they are eligible to continue, they will continue taking vismodeib daily as before for another 7 weeks while they receive radiation therapy.
  Other Names: Erivedge
Radiation: Radiation therapy — Radiation therapy will be started after the patient has finished taking vismodegib for 12 weeks. They will receive radiation once a day, Monday through Friday, for 7 weeks. Each radiation treatment may take up to 30 minutes.

SUMMARY:
Chemotherapy, radiation therapy, and surgery are standard treatments for basal cell carcinoma at most institutions. The purpose of this study is to determine whether adding vismodegib to radiation (chemoradiotherapy) is safe and tolerable. The purpose of this study is to assess the safety and tolerability of combined radiation therapy and vismodegib. This combination may increase the chances of the tumors being destroyed or unable to spread to other parts of the body in people with locally advanced basal cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
This is a single arm, multi-center Phase II clinical trial to assess the safety and demonstrate the efficacy of a combined modality approach using radiation therapy after induction and concurrently with systemic administration of vismodegib, which may increase the rates of complete response and sustained local control in patients with locally advanced Basal Cell Carcinoma (BCC)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced BCC of the head and neck, consisting of at least one histologically or cytologically confirmed lesion greater than or equal to 20 mm in longest diameter that is considered to be inoperable or to have a medical contraindication to surgery, in the opinion of a Mohs dermatologic surgeon, head and neck surgeon, or plastic surgeon. Locally advanced disease is considered to include involved lymph nodes of the neck. A patient with regionally involved lymph nodes in the neck is considered eligible. The patient should be considered a candidate for radiotherapy and should not have medical contraindications to receipt of radiation therapy.

   If a patient has distant metastatic spread of BCC (e.g., spread to distant areas outside the regional lymph nodes, clearly non contiguous areas of bone involvement, or distant metastasis to lung, brain, or other visceral organs), the patient should be considered as having distant metastasis and is not eligible.

   Note: All lesions that the investigator proposes to follow as target lesions during the course of the study must have previously been histologically confirmed as BCC.

   Acceptable contraindications to surgery include:
   * BCC that has recurred in the same location after two or more surgical procedures and successful curative resection is deemed unlikely
   * Complete surgical resection is not possible or is deemed excessively morbid (e.g. invasion into cranial nerves or skull base, proximity to brain, spinal canal, or orbit)
   * Anticipated substantial morbidity and/or major deformity from surgery (e.g. removal of a major facial structure, such as nose, ear, eyelid, eye, or jaw; or requirement for upper limb amputation)
   * Medical contraindication to surgery
   * Patient refusal of surgery due to anticipated morbidity
   * Other conditions considered to be contraindicating must be discussed with Data Coordinator before enrolling the patient.
2. Prior radiation therapy is acceptable but there cannot be major overlap of the previously irradiated tissues with the new radiation treatment volumes anticipated to be delivered for the purposes of this protocol, in such a way that curative intent with radiation cannot be met. Furthermore, the total dose from all radiation delivered and expected to be delivered should not exceed the suggested dose constraints given for normal structures.
3. Zubrod Performance Status 0-2
4. Age of greater than or equal to 18 years
5. Adequate bone marrow and organ function defined as follows:

   Adequate bone marrow function:

   leukocytes:> 3,000/microliter (mcL) absolute neutrophil count: greater than or equal to 1000 cells/mm3 platelets: greater than or equal to 75,000 cells/mm3 hemoglobin: greater than or equal to 8.5 g/dl (recommended cutoff subject to judgment of medical oncologist), but cannot be transfusion dependent

   Adequate hepatic function:

   total bilirubin: less than or equal to 1.5x institutional upper limit of normal (ULN) or within 3x the ULN for patients with Gilbert disease aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) : < 3 X institutional upper limit of normal alanine aminotransferase (ALT) /serum glutamic-pyruvic transaminase (SGPT): < 3 X institutional upper limit of normal

   Adequate renal function:

   creatinine: within normal institutional limits OR creatinine clearance: > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
6. Agreement not to donate blood or blood products during the study and for 7 months after discontinuation of vismodegib; for male patients, agreement not to donate sperm during the study and for 7 months after discontinuation of vismodegib.
7. For male patients, agreement not to donate sperm during the study and for 3 months after the final dose of vismodegib. Male patients must use condoms at all times, even after a vasectomy, during sexual intercourse with pregnant partners or female partners of reproductive potential during treatment with vismodegib. Vismodegib is present in semen. It is not known if the amount of vismodegib in semen can cause embryo-fetal harm.
8. Verify the pregnancy status of females of reproductive potential within 7 days prior to initiating vismodegib. For women of childbearing potential, a negative pregnancy test within 7 days prior to commencement of dosing is required. Women of reproductive potential are required to use two forms of acceptable contraception (including one acceptable barrier method with spermicide) during therapy and for 7 months after completing therapy. Acceptable forms of primary contraception include the following: Combination hormonal contraceptives, subcutaneous hormonal implant, hormonal patch, hormonal contraceptives (levonorgestre-releasing intrauterine system, medroxyprogesterone acetate depot), tubal sterilization, vasectomy, and intrauterine device (IUD). Acceptable forms of barrier contraception include the following: any male condom (with spermicide) or diaphragm (with spermicide).

Exclusion Criteria:

1. Patients with distant metastasis (e.g. spread to distant areas outside the regional lymph nodes, clearly non contiguous areas of bone involvement, or distant metastasis to lung, brain, liver or other visceral organs) are ineligible.
2. Patients with nevoid BCC syndrome (Gorlin syndrome) should not enroll in this study.
3. A patient with a known other malignancy is eligible if there is a negligible risk for disease progression or death within one year, there is no active ongoing treatment for this malignancy, and the malignancy and/or any anticipated future treatments would not interfere with protocol-mandated evaluations at 1 year.
4. Prior vismodegib or other antagonists of the Hh pathway;
5. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy, topical therapy such as 5-Fluorouracil or imiquimod, radiation therapy, surgery, or photodynamic therapy.

   * For patients with multiple cutaneous BCCs at baseline that are not designated by the investigator as target lesions, treatment of these non-target BCCs with surgery may be permitted but must be discussed with Data Coordinator prior to any surgical procedure.
6. Recent (within 4 weeks of Registration), current, or planned participation in another experimental drug study.
7. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields in such a way that curative intent with radiation cannot be met
8. Inability or unwillingness to swallow capsules; Patients with any condition that may impair the ability to swallow or absorb oral medications/investigational product including:

   * any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow capsules or pills;
   * prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel;
   * active peptic ulcer disease;
   * malabsorption syndrome
9. Pregnant or lactating women. Patients who are unable or are unwilling to adhere to the required contraceptive methods are excluded from the study.

   * Women of reproductive potential are required to use two forms of acceptable contraception (including one acceptable barrier method with spermicide) during therapy and for 7 months after completing therapy. Acceptable forms of primary contraception include the following: Combination hormonal contraceptives, subcutaneous hormonal implant, hormonal patch, hormonal contraceptives (levonorgestre-releasing intrauterine system, medroxyprogesterone acetate depot), tubal sterilisation, vasectomy and intrauterine device (IUD). Acceptable forms of barrier contraception include the following: Any male condom (with spermicide) or diaphragm (with spermicide).
   * Male patients must use condoms at all times, even after a vasectomy, during sexual intercourse with female partners of reproductive potential during treatment with vismodegib and for 2 months after the last dose to avoid exposing a pregnant partner and unborn fetus to vismodegib.
10. Life expectancy of <1 year
11. Patients with widespread superficial multifocal BCC who are considered unresectable due to breadth of involvement and do not have a single definable area of disease amenable to radiation therapy targeting.

    Note: If an area including one or more lesions is definable for radiation therapy targeting, the patient may be eligible for treatment on study using the designated target lesion(s) identified by the investigator.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements;
13. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk form treatment complications
14. HIV-positive patients on combination antiretroviral therapy, because of the potential for pharmacokinetic interactions with vismodegib;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vismodegib and Radiation Therapy: 150mg Vismodegib will be taken once a day, daily. Radiation therapy will be started after the patient has completed taking vismodegib for 12 weeks. The patient will take daily vismodegib through the completion of radiation therapy. The patient will receive radiation once a day, Monday through Friday, for 7 weeks. Each radiation treatment may take up to 30 minutes. After 12 weeks, they will be evaluated again to make sure they are still eligible to participate in the study. If they are eligible to continue, they will continue taking vismodeib daily as before for another 7 weeks while they receive radiation therapy.
Period: Overall Study
Arm/Group | Vismodegib and Radiation Therapy
Started | 24
Completed | 17
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 5
  60-69 years old | 8
  70-79 years old | 4
  80-89 years old | 6
  90-99 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Local-regional Control Rate
Description: The local-regional control rate at 12 months from protocol therapy completion, defined as absence of progressive disease within the irradiated planning tumor volumes (PTV) for patients with locally advanced basal cell carcinoma in the head and neck.
Time Frame: Up to 12 months after completing therapy
Measure: Number; unit: percentage
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
percentage | 100

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Estimate of the probability of PFS, with failure defined as any disease recurrence or death due to any cause with each duration measured from the time of first treatment with vismodegib to 12 months after completion of study treatment
Time Frame: From treatment start up to 12 months after completing therapy
Measure: Number; unit: probability of progression-free survival
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
probability of progression-free survival | 1.00

3. Secondary Outcome: Overall Survival (OS)
Description: Estimate of the probability of OS, with failure defined as any disease recurrence or death due to any cause with each duration measured from the time of first treatment with vismodegib to 12 months after completion of study treatment
Time Frame: From treatment start up to 12 months after completing therapy
Measure: Number; unit: probability of survival
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
probability of survival | 1.00

4. Secondary Outcome: Percentage of Patients by Treatment-Related Adverse Events by Event Description
Description: The percentage of any adverse events (CTCAE, v. 4.0) assessed to be definitely, probably, or possibly related to vismodegib or its combination with radiation therapy at any point during protocol therapy or during the followup period.
Time Frame: up to 12 months after completing therapy
Measure: Number; unit: percentage of patients
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 24
percentage of patients
  Grade 4 eye disorder | 4
  Grade 3 hyponatremia | 13
  Grade 3 oral mucositis | 8
  Grade 3 Gastrointestinal disorder | 8
  Grade 3 Dermatologic disorder | 8
  Grade 3 Abnormal Liver function | 4
  Grade 3 Anemia | 4
  Grade 3 Hypertension | 4
  Grade 2 Dermatitis | 33
  Grade 2 Dysgeusia | 33
  Grade 2 Myalgia | 25
  Grade 2 Fatigue | 21
  Grade 2 Oral mucositis | 21
  Grade 2 Weight Loss | 17

5. Secondary Outcome: Percentage of Patients by Adverse Event Not Related to Disease Progression
Description: The percentage of patients experiencing Grade 4-5 adverse events classified using CTCAE v.4.1 assessed to be definitely, probably, or possibly related to the induction or concurrent treatment components of the protocol regimen (that is not definitely related to disease progression) at any point during protocol therapy or during the followup period
Time Frame: up to 12 months after completing therapy
Population: Only 1 patient experienced an adverse event (Grade 4 Eye Disorder) not related to disease progression
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
percentage of participants | 6

6. Secondary Outcome: Number of Patients Discontinuing Treatment Due to Toxicity
Description: Feasibility of administering concurrent vismodegib with radiation therapy was assessed by the number of patients discontinuing treatment due to toxicity during the concurrent administration of vismodegib and radiation therapy (<75% of planned radiation therapy delivered)
Time Frame: up to 6 months from treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 24
Participants | 5

7. Secondary Outcome: Clinical Response Rate
Description: Response rate (as per RECIST) of the primary site and regionally involved areas following all treatment components at 3 months after the completion of protocol therapy will be reported as a percentage of the total sample.
Time Frame: Up to 12 months after completing therapy
Measure: Number; unit: percentage of patients
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
percentage of patients | 88

8. Secondary Outcome: Percentage of Patients With a Decrease of Basal Cell Carcinoma (BCC)
Description: Proportion of patients with a decrease of BCC within the irradiated planning tumor volumes (PTV) in patients who complete initial combined therapy, indicating a clinical response to vismodegib and radiation therapy
Time Frame: Up to 12 months after completing therapy
Measure: Number; unit: percentage of patients
Arm/Group | Vismodegib and Radiation Therapy
Number analyzed (Participants) | 17
percentage of patients | 88

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Vismodegib and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib and Radiation Therapy (N=24)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Corneal ulcer (Eye disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Abdominal Aortic Aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib and Radiation Therapy (N=24)
Dysgeusia (Nervous system disorders) | 19 (30)
Headache (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Dizziness (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (22)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 19 (26)
General disorders and administration site conditions - other (General disorders) | 4 (12)
Edema face (General disorders) | 2 (2)
Facial pain (General disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 8 (16)
Dry mouth (Gastrointestinal disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 10 (13)
Alanine aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 11 (18)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT01835626/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT01835626/ICF_001.pdf